CLINICAL TRIAL: NCT03718637
Title: Efficacy Evaluation of Surgical Treatment Using Bioinductive Implant for Tennis Elbow (Lateral Epicondylitis)
Brief Title: Efficacy Bioinductive Implant for Tennis Elbow (Lateral Epicondylitis)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Stephanie Muh, MD, Deputy Service Chief, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12495
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: Tennis Elbow; Tendinopathy; Lateral Epicondylitis; Bioinductive
MeSH Terms: conditions — Tennis Elbow; Tendinopathy | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups. In the "control group," patients will receive the current surgical treatment for lateral epicondylitis: tendon debridement and repair. Patients in the "experimental group" will receive a bio-inductive patch following the same surgical treatment. Both groups of patients will participate in preoperative and postoperative ultrasound imaging studies.
Who Masked: Participant
Masking Description: The study participant will not have knowledge of which treatment group he/she is randomized into for the duration of the study. Because the care provider/investigator will be required to implant the bioinductive patch, the physician will know into which treatment group each patient falls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Surgical treatment alone, consisting of tendon debridement and repair. Ultrasounds preoperatively and 6 months postoperatively.
  Interventions: Procedure: Lateral Epicondylectomy; Radiation: Ultrasound Imaging
- Experimental (Experimental): Identical surgical treatment plus Smith & Nephew bio-inductive patch implant. Ultrasounds preoperatively and 6 months postoperatively.
  Interventions: Biological: Smith & Nephew Bioinductive Implant; Procedure: Lateral Epicondylectomy; Radiation: Ultrasound Imaging

INTERVENTIONS:
Biological: Smith & Nephew Bioinductive Implant — A bioinductive implant that is supposed to foster healthy tendon regrowth after surgery.
  Other Names: Bioinductive Patch
  Arms: Experimental
Procedure: Lateral Epicondylectomy — This procedure is the standard of care for lateral epicondylitis patients who fail conservative treatment options.
Radiation: Ultrasound Imaging — An ultrasound will be performed on each patient both preoperatively and at 6 months.

SUMMARY:
The investigators are testing the efficacy of a new, FDA-approved bioinductive patch in lateral epicondylitis (tennis elbow) patients. A bioinductive patch is an implant that may foster tendon regrowth and healing following surgery. Patients will be randomize into one of two groups: control and investigational. Patients in the "control group" will receive the normal surgery for patients who do not respond to physical therapy, lifestyle changes, and anti-inflammatory treatment. Patients in the "experimental group" will receive the same surgical treatment, with the addition of the bioinductive patch. This patch will be implanted during surgery. Then, using a combination of ultrasound studies and other measures, the investigators will assess how well the patch works compared to surgery alone.

DETAILED DESCRIPTION:
A bioinductive patch is an implant that may foster tendon regrowth and healing following surgery. Patients will be randomized into one of two groups: control and investigational. All surgical patients will have failed non surgery options for 6 months (physical therapy, lifestyle changes, anti-inflammatories, injections) Patients in the "control group" will receive the standard surgery (open lateral epicondylectomy) . Patients in the "experimental group" will receive the same surgical treatment, with the addition of the bioinductive patch. This patch will be implanted during surgery. Then, using a combination of ultrasound studies and other measures, the investigators will assess how well the patch works compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lateral epicondylitis (tennis elbow) that has failed conservative treatment (Physical therapy, activity change, anti-inflammatory treatment.

Exclusion Criteria:

* Previous surgery on the currently-affected elbow.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
PROMIS CAT Scores | Preoperative to 1 year postoperative
  A short 5 minute survey asking questions about physical function, pain, and mental health
Visual Analog Scale (VAS) for Pain | Preoperative to 1 year postoperative
  Traditional 1 to 10, subjective rating of pain the patient is experiencing
Range of Motion | Preoperative to 1 year
  Standard range of motion values collected by the surgeon during preoperative and followup visits

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Muh, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.